CLINICAL TRIAL: NCT05602389
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Assess the Effect of Multi-herb Formulae VL-G-A57 and an Ashwagandha Root Formula (VL-G-E12) on the Modulation of the Hypothalamic-pituitary-adrenal Axis (HPA Axis) and Related Symptoms
Brief Title: Study to Assess the Effect of Multi-herb Formulae and an Ashwagandha Root Formula on the Modulation of the Stress and Related Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GH/220602/A57E12/HPA
Record Dates: First submitted 2022-10-21; First posted 2022-11-02 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Stress

STUDY DESIGN:
Intervention Model Description: Study Products: VL-G-A57 (Arm 1), VL-G-E12 (Arm 2) & Placebo (Arm 3) Dose: 700 mg daily Route: Oral Regimen: 2 capsules in the morning with food and 2 capsules in the evening with food Duration: 60 days
Who Masked: Participant, Investigator
Masking Description: A randomized, placebo-controlled, double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VL-G-A57 (Experimental): Dose: 700mg daily Route: Oral Regimen: 2 capsules in the morning with food and 2 capsules in the evening with food Duration: 60 days
  Interventions: Other: VL-G-A57
- VL-G-E12 (Experimental): Dose: 700mg daily Route: Oral Regimen: 2 capsules in the morning with food and 2 capsules in the evening with food Duration: 60 days
  Interventions: Other: VL-G-E12
- Placebo (Placebo Comparator): Dose: 700mg daily Route: Oral Regimen: 2 capsules in the morning with food and 2 capsules in the evening with food Duration: 60 days
  Interventions: Other: Placebo

INTERVENTIONS:
Other: VL-G-A57 — Dose: 700mg daily Route: Oral Regimen: 2 capsules in the morning with food and 2 capsules in the evening with food Duration: 60 days
  Arms: VL-G-A57
Other: VL-G-E12 — Dose: 700mg daily Route: Oral Regimen: 2 capsules in the morning with food and 2 capsules in the evening with food Duration: 60 days
  Arms: VL-G-E12
Other: Placebo — Dose: 700mg daily Route: Oral Regimen: 2 capsules in the morning with food and 2 capsules in the evening with food Duration: 60 days
  Arms: Placebo

SUMMARY:
Two unique proprietary formulations of adaptogens VL-G-E12 formulation and an herbal blend containing VL-G-A57 is one of the most well-known adaptogens that has been used for years to enhance positive mood states, deepen sleep, and improve memory. The product has been proven to have a role in improving depression, enhancing work performance, eliminating fatigue and treating symptoms of asthenia subsequent to intense physical and psychological stress. The extract was tested on antidepressant, adaptogenic, anxiolytic, nociceptive and locomotor activities at doses of 10, 15 and 20 mg/kg, using predictive behavioral tests and animal models. The results show that this product extract significantly, but not dose-dependently, induced antidepressant-like, adaptogenic, anxiolytic-like and stimulating effects in mice. Studies reveal that this shrub has antimicrobial (including antibacterial, antiviral, antifungal, antiprotozoal, antimalarial, anthelmintic), anti-inflammatory, anti-diabetic, anti-hypercholesterolemia, anti-hypertensive, anti-carcinogenic, and immunomodulatory effect.The aim of the current study is to assess the adaptogenic effects of two potential investigational products VL-G-A57 and VL-G-E12 Their adaptogenic effect shall be investigated by assessing several clinical symptoms of HPA axis dysfunction such as stress, anxiety, sleep quality, fatigue, mood etc.

ELIGIBILITY:
Inclusion Criteria

1. Male and female subjects ≥18 and ≤ 65 years' old with active lifestyle, moderate physical activity level as per International Physical Activity Questionnaire - Short Form (IPAQ - SF)
2. BMI: 18 to 29.9 kg/m2
3. RSQ-W (Restorative Sleep Questionnaire-weekly version) score less than or equal to 50
4. PSS scores ranging from 27-40
5. All participants will be encouraged to not make any major lifestyle changes during the study period.
6. They will be informed that any major changes may result in exclusion from the study.
7. Participants willing to provide written informed consent.

Exclusion Criteria

1. Subjects with a medical history of heart disease, respiratory disorders, metabolic or lifestyle disorders, seizure disorders, or other chronic health conditions requiring medication were excluded.
2. Individuals who currently, or in the past 6 months suffered from any diagnosable mental-health disorder (as assessed by the Mini International Neuropsychiatric Interview 5.0.01 ) or were taking apsychotropic medication or other herbal preparation were also excluded from participating in the study.
3. Subjects with a blood pressure range of systolic ≥ 140 mm Hg and diastolic ≥ 90 mm Hg.
4. Subjects on any sleep medication since last 3 months
5. Subjects with a history of severe intrinsic sleep related disorders.
6. Subjects who have taken Ashwagandha or any sleep or other supplements within the last three months,
7. People with a known hypersensitivity to Ashwagandha
8. Subjects who work on a night shift
9. Nursing or pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Perceived stress scale | Day 0
  To assess the impact of the Investigational Product (IP) on stress levels by using the Perceived stress scale (PSS)from baseline.
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress.
Perceived stress scale | Day 30
  To assess the impact of the Investigational Product (IP) on stress levels by using the Perceived stress scale (PSS)from baseline.
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress.
Perceived stress scale | Day 60
  To assess the impact of the Investigational Product (IP) on stress levels by using the Perceived stress scale (PSS)from baseline.
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index. | Day 0, 30 and 60
  To assess sleep quality using Pittsburgh Sleep Quality Index.
  In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21).
  Higher scores indicate worse sleep quality.
Restorative sleep questionnaire | Day 0, 30 and 60
  To assess change in the total score of the restorative sleep questionnaire weekly RSQ-W is a validated scale for measuring refreshing quality of sleep. It has 9 items with answers scaled from 1 to 5. The questioned asked about one felt after waking up and starting the day during the past seven days. Refer to the questionnaire at Appendix 3
  Question 9 is to be reversed scored. The total score is an average score based on all 9 items and rescaled to a 0 to 100 scale, using the following transformation:
  RSQ-W Total Score = (RSQ-W average score across completed items - 1) X 25. The participants will be asked to administer this scale during screening visit. Those fulfilling the criteria (RSQ-W score ≤ 50), will further fill this scale at day 0, day 30 and day 60 for assessing the efficacy.
Adrenocorticotropic Hormone (ACTH) in plasma | Day 0, 30 and 60
  To assess changes in Adrenocorticotropic Hormone (ACTH) in plasma
Morning Salivary Cortisol | Day 0, 30 and 60
  To assess changes in morning Salivary Cortisol
Impact of the IP on the Mental alertness | Day 0, 30 and 60
  To assess the impact of the IP on the Mental alertness of the participants using a three-pointer scale after rising The scoring will be done as following: 1 = alert, 2 = slightly drowsy and 3 = extremely drowsy
Fatigue Severity Scale | Day 0, 30 and 60
  To assess the impact of IP on Fatigue using the Fatigue Severity Scale. The FSS is a self-administered questionnaire with 9 items (questions) investigating the severity of fatigue in different situations during the past week. Grading of each item ranges from 1 to 7, where 1 indicates strong disagreement and 7 indicates strong agreement, and the final score represents the mean value of the 9 items. A visual analogue scale is also included with the scale in which the respondents will be asked to denote the severity of their fatigue at the present moment by placing a mark on a line extending from "no fatigue" to "fatigue as bad as could be." Higher scores on the scale are indicative of more severe fatigue.
Depression, Anxiety, Stress Scale-21 | Day 0, 30 and 60
  To assess the impact of the IP on total scores of Depression, Anxiety, Stress Scale-21 Higher score indicates worst Depression, Anxiety, Stress.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shalini Srivastava, MD medicine, Principal Investigator — Vedic Lifesciences Pvt. Ltd.
Locations (5):
- India (5):
  - Vedic Lifesciences PVT LTD, Mumbai, Maharashtra
  - Stress test clinic, Mumbai, Maharashtra
  - Shree Polyclinic, Mumbai, Maharashtra
  - The Kewalramani Clini, Mumbai, Maharashtra
  - Dr Chandrakant Mishra clinic, Pālghar, Maharashtra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McKinney E, Stewart J, Kewalramani R, Singh S. Effects of multi-herb and ashwagandha root formulas on stress modulation: a randomized, double-blind, placebo-controlled clinical study. Trials. 2026 Feb 9. doi: 10.1186/s13063-026-09495-9. Online ahead of print. PMID 41656269